CLINICAL TRIAL: NCT06579833
Title: Histotripsy (HistoSonics®) for Liver Tumours: a Phase II Safety and Efficacy Study
Brief Title: Histotripsy (HistoSonics®) for Liver Tumours
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Albert Chi Yan Chan, Clinical Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW24-442
Record Dates: First submitted 2024-08-13; First posted 2024-08-30 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Liver Tumour
Keywords: liver tumour
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Histotripsy (Other): Histotripsy is a promising non-invasive technique that uses high-intensity ultrasound waves to disrupt tissue without damaging surrounding structures
  Interventions: Radiation: Histotripsy

INTERVENTIONS:
Radiation: Histotripsy — Histotripsy is a promising non-invasive technique that uses high-intensity ultrasound waves to disrupt tissue without damaging surrounding structures. It works by using high-intensity ultrasound waves to create microscopic bubbles within the tumour tissue. These bubbles rapidly expand and collapse, generating shock waves that disrupt the tissue. The technique is highly precise and can be targeted to specific areas of the liver, allowing for selective destruction of tumour cells while minimizing damage to healthy tissue.
  Other Names: HistoSonics

SUMMARY:
Histotripsy is a promising non-invasive technique that uses high-intensity ultrasound waves to disrupt tissue without damaging surrounding structures. It works by using high-intensity ultrasound waves to create microscopic bubbles within the tumour tissue. These bubbles rapidly expand and collapse, generating shock waves that disrupt the tissue. The technique is highly precise and can be targeted to specific areas of the liver, allowing for selective destruction of tumour cells while minimizing damage to healthy tissue. This study will enrol 20 patients with liver tumours (be it primary or secondary liver tumours), monitor their post-operative adverse events, and study the changes in tumour size and volume after treatment. Histotripsy will be performed under general anaesthesia, with real-time monitoring by ultrasound, and deliver high-intensity ultrasound waves in single session or multiple sessions. Similar to other minimal invasive treatments, patients will be admitted 1 day prior, then receive Histotripsy on the next day and stay overnight for observation. Patients will be discharged on the 3rd day if unremarkable. During the hospital stay, blood samplings will be taken for evaluation around 2-4 times in total depending on the length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Fit for general anaesthesia
* Liver tumour size < 10cm
* Solitary or multifocal
* Primary liver tumour such as hepatocellular carcinoma or intrahepatic cholangiocarcinoma
* Secondary liver tumour such as liver metastasis
* Patients with operable or inoperable liver tumours
* Liver transplant candidates awaiting for liver graft

Exclusion Criteria:

* Refusal to take part in clinical trial
* Child C liver cirrhosis
* Not fit for general anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in tumour features | up to 36 months
  Changes in tumour size and volume before and after intervention
Post procedure adverse events and complication | The whole duration of hospital stay, normally 3 days on average
  Post procedure adverse events and complication

CONTACTS AND LOCATIONS:
Overall Officials: Albert Chan, MS, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No